CLINICAL TRIAL: NCT06031623
Title: Effect Of Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest (REBOA); A Multinational, Multicenter Randomized Controlled Trial
Brief Title: REBOA in Nontraumatic OHCA
Acronym: REBOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dong Keon Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Arrest
Keywords: Advanced cardiopulmonary resuscitation (ACLS); Cardiopulmonary resuscitation (CPR); Resuscitative endovascular balloon occlusion of the aorta (REBOA)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients allocated to this arm receives conventional resuscitative measures according to the 2020 AHA CPR Guidelines.
- REBOA (Experimental): After enrollment and randomization, patients allocated to this arm receives REBOA in addition to conventional ACLS according to the 2020 AHA CPR guidelines. The common femoral artery is accessed with ultrasound guidance. A sheath catheter is inserted, followed by a REBOA catheter. The REBOA is ballooned with 20cc of normal saline or until resistance is felt.
  Interventions: Device: REBOA

INTERVENTIONS:
Device: REBOA — Resuscitative endovascular balloon occlusion of the aorta (REBOA)is a device composed of a catheter attached to an inflatable balloon. It is inserted through the common femoral artery and guided to the thoracic aorta.
  Arms: REBOA

SUMMARY:
The investigators propose a multicenter randomized controlled trial in South Korea and Taiwan to observe the clinical effects of REBOA on nontraumatic out-of-hospital-cardiac-arrest (OHCA) patients. While REBOA has been traditionally used in trauma for hemorrhage control, it has also shown promising results in nontraumatic cardiac arrests by rerouting circulation to increase perfusion in the coronary and brain.

DETAILED DESCRIPTION:
Nontraumatic OHCA patients arriving at the 2 participating hospitals between the ages of 20 to 80 will be eligible. If the patient meets the enrollment criteria, he/she will be randomized into the control group (treatment with conventional ACLS according to the 2020 AHA guideline) or the REBOA group (ACLS according to the 2020 AHA guideline with REBOA application). A sheath catheter is inserted with ultrasound guidance to gain access to the common femoral artery in both groups. This is followed by insertion of the REBOA catheter, if the patient is allocated into the intervention group. The aortic balloon is inflated. If ROSC is achieved, the balloon is deflated slowly. Patients who achieve ROSC will receive post cardiac arrest management according to the 2020 AHA guideline.

ELIGIBILITY:
Inclusion Criteria:

* Adult nontraumatic OHCA
* Witnessed arrest
* Arrival at ER from 9AM to 5PM (in South Korea) and 8AM to 8PM (in Taiwan)

Exclusion Criteria:

1. age below 20 years old or over 80 years old,
2. traumatic cardiac arrest,
3. those with unwitnessed cardiac arrest,
4. pregnant patients,
5. patients who have already achieved ROSC upon arrival at the emergency department
6. pre-cardiac arrest cerebral performance category of 3-4
7. those showing evidence of cardiac arrest due to bleeding (such as gastrointestinal bleeding)
8. those suspected of having aortic disease, such as dissection, intramural hematoma, or aneurysm, by bedside ultrasound performed immediately after ED arrival or have a previous history of aortic disease
9. whose legal representative has requested termination of resuscitation efforts before study enrollment
10. declared dead at scene before randomization
11. Patients who meet the criteria for extracorporeal cardiopulmonary resuscitation (ECPR), and therefore the decision is made to perform ECPR, will not be enrolled. The ECPR criteria applies when all of the following criteria are met: pre-cardiac arrest CPC of 1-2, witnessed cardiac arrest with bystander CPR, ages between 20-70, initial shockable rhythm, ECMO pump-on available within 60 minutes of onset of cardiac arrest, and patients without end-stage diseases such as cancer, liver cirrhosis, or end-stage renal failure.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Achieved ROSC (return of spontaneous circulation) | 24 hours
  Number of patients who achieves ROSC regardless of sustained time

SECONDARY OUTCOMES:
Number of Participants Who Achieved Sustained ROSC | 24 hours
  Number of participants who achieves sustained ROSC (ROSC maintained more than 20 minutes)
Survival to Admission | 48 hours
  Whether patients who achieve sustained ROSC survives until admission
Survival to Discharge | 30 days
  Whether patients survive until hospital discharge.
Neurological Outcome | 1 month, 3 months, 6 months since ROSC
  The cerebral performance category (CPC) and modified Rankin Score (mRS) of each patient at 28 days, 3 months, and 6 months after achieving ROSC. CPC is measured on a scale of 1 to 5, with 1 being the best neurological performance, and 5 indicating brain death. MRS is measured on a scale of 0 to 6, with 0 indicating no neurological deficit, and 6 indicating death.
Changes in Arterial Blood Pressure | ABP 2 minutes and 1 minute before REBOA insertion, ABP 1 minute / 2 minutes / 4 minutes / 10 minutes after REBOA insertion.
  Arterial blood pressure measured before and after REBOA inflation in the experimental group. Both systolic and diastolic pressures will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univeristy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang DH, Lee DK, Jo YH, Park SM, Oh YT, Im CW. Resuscitative endovascular occlusion of the aorta (REBOA) as a mechanical method for increasing the coronary perfusion pressure in non-traumatic out-of-hospital cardiac arrest patients. Resuscitation. 2022 Oct;179:277-284. doi: 10.1016/j.resuscitation.2022.07.020. Epub 2022 Jul 21. PMID 35870557
- [Background] Brede JR, Lafrenz T, Klepstad P, Skjaerseth EA, Nordseth T, Sovik E, Kruger AJ. Feasibility of Pre-Hospital Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2019 Nov 19;8(22):e014394. doi: 10.1161/JAHA.119.014394. Epub 2019 Nov 11. PMID 31707942
- [Background] Mazzoli CA, Chiarini V, Coniglio C, Lupi C, Tartaglione M, Gamberini L, Semeraro F, Gordini G. Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in Non-Traumatic Cardiac Arrest: A Narrative Review of Known and Potential Physiological Effects. J Clin Med. 2022 Jan 29;11(3):742. doi: 10.3390/jcm11030742. PMID 35160193
- [Background] Daley J, Morrison JJ, Sather J, Hile L. The role of resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to ACLS in non-traumatic cardiac arrest. Am J Emerg Med. 2017 May;35(5):731-736. doi: 10.1016/j.ajem.2017.01.010. Epub 2017 Jan 12. PMID 28117180
- [Background] Nowadly CD, Johnson MA, Hoareau GL, Manning JE, Daley JI. The use of resuscitative endovascular balloon occlusion of the aorta (REBOA) for non-traumatic cardiac arrest: A review. J Am Coll Emerg Physicians Open. 2020 Aug 30;1(5):737-743. doi: 10.1002/emp2.12241. eCollection 2020 Oct. PMID 33145513
- [Background] Hutin A, Levy Y, Lidouren F, Kohlhauer M, Carli P, Ghaleh B, Lamhaut L, Tissier R. Resuscitative endovascular balloon occlusion of the aorta vs epinephrine in the treatment of non-traumatic cardiac arrest in swine. Ann Intensive Care. 2021 May 17;11(1):81. doi: 10.1186/s13613-021-00871-z. PMID 34002305
- [Derived] Kim HE, Chu SE, Jo YH, Chiang WC, Jang DH, Chang CH, Oh SH, Chen HA, Park SM, Sun JT, Lee DK. Effect of resuscitative endovascular balloon occlusion of the aorta in nontraumatic out-of-hospital cardiac arrest: a multinational, multicenter, randomized, controlled trial. Trials. 2024 Feb 13;25(1):118. doi: 10.1186/s13063-024-07928-x. PMID 38347550

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT06031623/Prot_SAP_ICF_003.pdf